CLINICAL TRIAL: NCT06983236
Title: Exploring Nursing Students' Ability to Create Artificial Intelligence-Enhanced Patient Education Materials on Infection Care: A Randomized Controlled Trial
Brief Title: Exploring Nursing Students' Ability to Create Artificial Intelligence-Enhanced Patient Education Materials on Infection Care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Gülsüm Çonoğlu, Dr. Lecturer, Çankırı Karatekin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 5064223087
Record Dates: First submitted 2025-05-05; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Nursing Students; Artificial Intelligence (AI); Patient Education Materials; Randomized Controlled Trial
Keywords: Nursing Students; Artificial Intelligence (AI); Patient Education Materials; Randomized controlled trial

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Students in the intervention group will be asked to prepare patient education material for a patient using an artificial intelligence (AI) tool on 'infection care'. First, the intervention group will receive 2 hours of training on artificial intelligence. This training will take place in a classroom environment with internet access. All students in the intervention group will be trained at the same time and their questions will be answered. The students will not receive any additional counselling after the training. It will be explained to the students in the intervention group that they will first have to prepare the educational material using the AI tool and that they can use support tools such as books, magazines and websites while preparing the educational material. Students will be given five days and will be asked to submit their patient education materials at the end of the five days and will be asked to complete the patient education information form.
  Interventions: Behavioral: AI-enabled patient education material
- Control group (Active Comparator): Students in the control group will be interviewed and asked to prepare a patient education material about "infection care" for a patient. Students will be informed that they can use additional tools such as books, magazines, and websites to prepare educational materials. Students will be given five days and at the end of the five days, they will be asked to submit their patient education materials and fill out the Patient Education Information Form. Students will be asked to write down the references they used in detail and include direct links to the websites of the Internet resources.
  Interventions: Behavioral: Traditional patient education material

INTERVENTIONS:
Behavioral: AI-enabled patient education material — Students in the intervention group will be asked to prepare patient education material for a patient using an artificial intelligence (AI) tool on 'infection care'. First, the intervention group will receive 2 hours of training on artificial intelligence. This training will take place in a classroom environment with internet access. All students in the intervention group will be trained at the same time and their questions will be answered. The students will not receive any additional counselling after the training. It will be explained to the students in the intervention group that they will first have to prepare the educational material using the AI tool and that they can use support tools such as books, magazines and websites while preparing the educational material. Students will be given five days and will be asked to submit their patient education materials at the end of the five days and will be asked to complete the patient education information form.
  Arms: Intervention group
Behavioral: Traditional patient education material — Students in the control group will be interviewed and asked to prepare a patient education material about "infection care" for a patient. Students will be informed that they can use additional tools such as books, magazines, and websites to prepare educational materials. Students will be given five days and at the end of the five days, they will be asked to submit their patient education materials and fill out the Patient Education Information Form. Students will be asked to write down the references they used in detail and include direct links to the websites of the Internet resources.
  Arms: Control group

SUMMARY:
The purpose of this study is to explore the ability of nursing students to create artificial intelligence-supported patient education materials regarding infection care. This study will be conducted as a randomized controlled experimental study. Data of the study will be collected with the Descriptive Characteristics Form, Patient Education Information Form and Patient Education Materials Assessment Tool (HEMDA).

ELIGIBILITY:
Inclusion Criteria:

* To take Basic Principles and Practices in Nursing-II for the first time
* Not to work as a nurse in a hospital or any health institution

Exclusion Criteria:

* Having previously prepared patient education materials;
* Retaking the Basic Principles and Practices in Nursing-II course
* Having difficulty speaking and understanding Turkish;
* Not attending class

Ages: 18 Years to 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-05-16 (Estimated); Primary Completion 2025-05-21 (Estimated); Study Completion 2025-06-25 (Estimated)

PRIMARY OUTCOMES:
Patient Education Information Form | day 6 after the intervention
  The form, prepared by researchers in line with the literature (Bastable, 2021; Orgun et al., 2024; Saatçi et al., 2024); includes questions regarding the subject of patient education, the tools/materials used in preparing patient education, the total time spent preparing patient education material, the resources used in patient education, and the level of satisfaction with the material preparation process.

SECONDARY OUTCOMES:
Patient Education Materials Assessment Tool (PEMAT-TR) | After the intervention from day 6 to 1 month after intervention
  The Turkish adaptation of the Patient Education Materials Assessment Tool (PEMAT), developed by Shoemaker, Wolf and Brach in 2014 to evaluate the understandability and applicability of printed/printable and audiovisual patient education materials, was made by Paylan Akkoç and Orgun (2023). There are two versions: "Patient Education Materials Assessment Tool for Printable Materials (PEMAT TR-P)" and "Patient Education Materials Assessment Tool for Audio-Visual Material (PEMAT TR-A/V)". The one to be used in this study is PEMAT TR-P, which consists of two dimensions: understandability (17 items) and applicability (7 items). Cronbach's alpha coefficient is 0.901 for the Turkish version of the Patient Education Materials Assessment Tool for Printable Materials. Each item in the scale is evaluated by giving a score of 0 (disagree) and 1 (agree), and there is a third option for the material as "No Evaluation (DA)" for some items.

IPD SHARING:
Plan to Share IPD: No
For ethical reasons